CLINICAL TRIAL: NCT05257824
Title: Optimal Duration of Dual Antiplatelet Therapy After Stent-assisted Coiling of Unruptured Intracranial Aneurysms: A Prospective Randomized Multicenter Trial
Brief Title: Optimal Duration of Dual Antiplatelet Therapy After Stent-assisted Coiling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Pusan National University Yangsan Hospital (Other); Keimyung University Dongsan Medical Center (Other); Uijeongbu St. Mary's Hospital (Unknown); Chungnam National University Sejong Hospital (Other); Soonchunhyang University Hospital (Other); Asan Medical Center (Other); Gangnam Severance Hospital, Yonsei University College of Medicine (Unknown)
Responsible Party: Principal Investigator, Kwon Oki, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-2102-667-002
Record Dates: First submitted 2022-02-11; First posted 2022-02-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aneurysm Cerebral; Endovascular Procedures
Keywords: dual antiplatelet; cerebral aneurysm; coil embolization; stent
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: 1. short-term dual antiplatelet group: for 6 months
  2. long-term dual antiplatelet group: for 12 months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- short-term dual antiplatelet group (Active Comparator): Patients with unruptured intracranial aneurysms received dual antiplatelet agents (100mg of aspirin and 75mg of clopidogrel) for at least five days before coil embolization. One day prior to coiling, aspirin reaction units (ARU) and P2Y12 reaction units (PRU) were measured using VerifyNow. Patients with proper aspirin and clopidogrel reaction units (ARU < 550 and PRU 85 ~219) will be enrolled in this study. After stent-assisted coiling, dual antiplatelet treatment continued for 6 months; after that time, this therapy will be exchanged for daily oral 100mg of aspirin for 18 months after coiling
  Interventions: Drug: Aspirin 100mg; Drug: Clopidogrel 75mg
- long-term dual antiplatelet group (Experimental): Patients with unruptured intracranial aneurysms received dual antiplatelet agents (100mg of aspirin and 75mg of clopidogrel) for at least five days before coil embolization. One day prior to coiling, aspirin reaction units (ARU) and P2Y12 reaction units (PRU) were measured using VerifyNow. Patients with proper aspirin and clopidogrel reaction units (ARU < 550 and PRU 85 ~219) will be enrolled in this study. After stent-assisted coiling, dual antiplatelet treatment continued for 12 months; after that time, this therapy will be exchanged for daily oral 100mg of aspirin for 18 months after coiling.
  Interventions: Drug: Aspirin 100mg; Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Aspirin 100mg — 1. short-term dual antiplatelet: dual antiplatelet agents for 6 months
  2. long-term dual antiplatelet: dual antiplatelet agents for 12 months
  Other Names: Aspirin protect; Aspirin enteric coated
Drug: Clopidogrel 75mg — 1. short-term dual antiplatelet: dual antiplatelet agents for 6 months
  2. long-term dual antiplatelet: dual antiplatelet agents for 12 months
  Other Names: Plavix; Celavix; Plavitor; Pregrel; Cloart; Platless; Pidogle; Antipla; Jgrel

SUMMARY:
Comparison of duration of dual antiplatelet therapy after stent-assisted coiling of unruptured intracranial aneurysms

DETAILED DESCRIPTION:
The purpose of this study is to compare the incidence of thromboembolic and hemorrhagic complications between 1 and 18 months after stent-assisted coiling according to the duration of use of dual antiplatelet agents (6 months versus 12 months) after stent-assisted coiling of unruptured intracranial aneurysms to determine the optimal duration of use of dual antiplatelet agents.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 19 years old
* subjects with modified Rankin Scale (mRS) ≤ 2
* subjects with unruptured intracranial aneurysms
* subjects with appropriated aspirin and clopidogrel reaction units after dual antiplatelet preparation (100 mg of aspirin and 75 mg of clopidogrel) for at least 5 days before procedure [measured using VerifyNow]

  1. aspirin reaction unit (ARU) < 550
  2. P2Y12 reaction unit (PRU): 85~219
* subjects who agreed to this study (with informed consent)

Exclusion Criteria:

* subjects with neurological deficits (mRS ≥ 3)
* subjects with an allergic reaction to antiplatelets (aspirin and clopidogrel) or contrast
* subjects with a high risk of hemorrhage such ICH or severe gastric ulceration
* subjects with coagulopathy
* subjects with thrombocytopenia (<100,000/mm3)
* subjects with liver diseases (> 100IU/L of aspartate aminotransferase or alanine aminotransferase)
* subjects with renal diseases (> 2mg/dL of serum creatinine)
* subjects with underlying diseases that need to maintain dual antiplatelet drugs or anticoagulants.
* subjects with a high risk of strokes (atrial fibrillation, over 70% cerebral artery stenosis or cerebral artery occlusion, moyamoya disease, vascular malformations, etc)
* subjects with uncontrolled congestive heart failure or angina
* subjects with malignant tumors
* subjects with a positive pregnancy test (serum or urine)
* subjects who are unconscious at the time of diagnosis.
* subjects who are unable to complete the required follow-ups
* subjects with life-threatening diseases
* subjects with medical conditions with a life expectancy of less than two years
* subjects who are determined to be disqualified by researchers

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-12-02 (Actual); Study Completion 2025-12-02 (Actual)

PRIMARY OUTCOMES:
Incidence of thromboembolic complications | between 1 and 18 months after stent-assisted coil embolization
  The primary outcome measure is incidence of thromboembolic complications between 1 and 18 months post-procedure.

SECONDARY OUTCOMES:
Incidence of periprocedural complications | during procedure and within 1 month post-procedure
  Incidence of periprocedural complications during procedure and within 1 month post-procedure
Incidence of hemorrhagic complications | between 1 and 18 months after stent-assisted coil embolization
  Incidence of hemorrhagic complications between 1 and 18 months post-procedure.
Changes of modified Rankin scale in clinical and functional outcomes at 18 months follow up | within 18 months post-procedure
  Changes in clinical and functional outcomes at 18 months follow up, as measured by an increase in the modified Rankin Scale compared to baseline (modified Rankin Scale: 0) no symptoms, 1) able to carry out all usual activities, despite some symptoms, 2) able to look after own affairs without assistance, but unable to carry out all previous activities, 3) requires some help, but able to wal unassisted, 4) unable to attend to own bodily needs without assistance, and unable to walk unassisted, 5) requires constant nursing care and attention, bedridden, incontinent and 6) dead.
Incidence of unrelated complication with this study | within 18 months post-procedure
  Incidence of myocardial infarction and unrelated thromboembolic or hemorrhagic complications with this study
Changes in aspirin reaction unit and P2Y12 reaction units at 6 months follow-up by using VerifyNow | at 6 months
  Change in aspirin reaction unit and P2Y12 reaction unit at the time of 6 months follow-up compared to baseline by using VerifyNow (Accumetrics, USA)
Periprocedural mortality | within 1 month
  Death within 1 month
Comparison of mortality | between 1 and 18 months after stent-assisted coil embolization
  Death between 1 and 18 months post-procedure
Changes in radiological outcomes by Roy-Raymond grades | at 18 months
  Change in radiological outcomes at 18 months follow up compared to baseline as measured by Roy-Raymond grades: 1) complete, 2) residual neck, and 3) residual sac

CONTACTS AND LOCATIONS:
Overall Officials: O-Ki Kwon, Principal Investigator — Seoul National University Bundang Hospital
Locations (8):
- South Korea (8):
  - Chungnam National University Sejong Hospital, Sejong, Chungcheongnam-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Soonchunhyang University Seoul Hospital, Seoul
  - Asan Medical Center, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Uijeongbu St. Mary's Hospital, Uijeongbu-si

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] UCAS Japan Investigators; Morita A, Kirino T, Hashi K, Aoki N, Fukuhara S, Hashimoto N, Nakayama T, Sakai M, Teramoto A, Tominari S, Yoshimoto T. The natural course of unruptured cerebral aneurysms in a Japanese cohort. N Engl J Med. 2012 Jun 28;366(26):2474-82. doi: 10.1056/NEJMoa1113260. PMID 22738097
- [Background] Hwang G, Kim JG, Song KS, Lee YJ, Villavicencio JB, Suroto NS, Park NM, Park SJ, Jeong EA, Kwon OK. Delayed ischemic stroke after stent-assisted coil placement in cerebral aneurysm: characteristics and optimal duration of preventative dual antiplatelet therapy. Radiology. 2014 Oct;273(1):194-201. doi: 10.1148/radiol.14140070. Epub 2014 Jun 11. PMID 24918960
- [Background] Hwang G, Huh W, Lee JS, Villavicencio JB, Villamor RB Jr, Ahn SY, Kim J, Chang JY, Park SJ, Park NM, Jeong EA, Kwon OK. Standard vs Modified Antiplatelet Preparation for Preventing Thromboembolic Events in Patients With High On-Treatment Platelet Reactivity Undergoing Coil Embolization for an Unruptured Intracranial Aneurysm: A Randomized Clinical Trial. JAMA Neurol. 2015 Jul;72(7):764-72. doi: 10.1001/jamaneurol.2015.0654. PMID 26010803
- [Background] Kim CH, Hwang G, Kwon OK, Ban SP, Chinh ND, Tjahjadi M, Oh CW, Bang JS, Kim T. P2Y12 Reaction Units Threshold for Implementing Modified Antiplatelet Preparation in Coil Embolization of Unruptured Aneurysms: A Prospective Validation Study. Radiology. 2017 Feb;282(2):542-551. doi: 10.1148/radiol.2016160542. Epub 2016 Sep 2. PMID 27603789
- [Background] Kim T, Kim CH, Kang SH, Ban SP, Kwon OK. Relevance of Antiplatelet Therapy Duration After Stent-Assisted Coil Embolization for Unruptured Intracranial Aneurysms. World Neurosurg. 2018 Aug;116:e699-e708. doi: 10.1016/j.wneu.2018.05.071. Epub 2018 May 17. PMID 29778598
- [Background] Hwang G, Jung C, Park SQ, Kang HS, Lee SH, Oh CW, Chung YS, Han MH, Kwon OK. Thromboembolic complications of elective coil embolization of unruptured aneurysms: the effect of oral antiplatelet preparation on periprocedural thromboembolic complication. Neurosurgery. 2010 Sep;67(3):743-8; discussion 748. doi: 10.1227/01.NEU.0000374770.09140.FB. PMID 20651627
- [Background] Almekhlafi MA, Al Sultan AS, Kuczynski AM, Brinjikji W, Menon BK, Hill MD, Goyal M. Antiplatelet therapy for prevention of thromboembolic complications in coiling-only procedures for unruptured brain aneurysms. J Neurointerv Surg. 2020 Mar;12(3):298-302. doi: 10.1136/neurintsurg-2019-015173. Epub 2019 Sep 20. PMID 31540948